CLINICAL TRIAL: NCT04507672
Title: Acetated Ringer's Solution Versus Saline in Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Zhongda Hospital,Southeast University, China, Southeast University, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018ZDSYLL105-P01
Record Dates: First submitted 2020-07-02; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Septic Shock Hyperdynamic
Keywords: Crystalloid; Renal failure; Renal dysfunction
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, multiple-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saline group (Placebo Comparator): Use saline for fluid resuscitation during the first 72 hours after enrollment
  Interventions: Drug: Fluid resuscitation
- Acetated Ringer's solution group (Experimental): Use acetated Ringer's solution for fluid resuscitation during the first 72 hours after enrollment
  Interventions: Drug: Fluid resuscitation

INTERVENTIONS:
Drug: Fluid resuscitation — Use the choice of crystalloid for resuscitation during the first 72 hours after enrollment

SUMMARY:
The primary aim of this trial is to compare the effect of acetated ringer's solution with that of saline for therapy on the incidence and development of major adverse renal events among septic shock patients. The investigators hypothesize that use of acetated ringer's solution for resuscitation among septic shock patients will reduce the incidence of major adverse kidney events.

DETAILED DESCRIPTION:
Normal saline and Ringer's solutions are the preferred crystalloid fluids administered in early septic shock. However, evidence have associated saline with hyperchloremia and secondary metabolic acidosis, and renal vasoconstriction, increased incidence of acute kidney injury (AKI) and mortality. The primary aim of this trial is to compare the effect of acetated ringer's solution with that of saline for therapy on the incidence and development of major adverse renal events among septic shock patients. The investigators hypothesize that use of acetated ringer's solution for resuscitation among septic shock patients will reduce the incidence of major adverse kidney events.

ELIGIBILITY:
Inclusion Criteria:

Adult patients presenting to the ICU diagnosed as septic shock within 24 hours.

Exclusion Criteria:

1. Pregnancy;
2. Likely requirement for immediate hemodialysis or renal replacement therapy;
3. Patients have already received fluids for more than 4 liters;
4. Patient in extremis or death deemed imminent and inevitable.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse renal events in 28 days | 28 day
  Incidence of major adverse renal events

SECONDARY OUTCOMES:
Incidence of kidney injury | 28 day
  Incidence of kidney injury
Serum creatinine（umol/L） | 28 day
  serum creatinine（umol/L）

REFERENCES:
- [Result] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Result] Peters E, Antonelli M, Wittebole X, Nanchal R, Francois B, Sakr Y, Vincent JL, Pickkers P. A worldwide multicentre evaluation of the influence of deterioration or improvement of acute kidney injury on clinical outcome in critically ill patients with and without sepsis at ICU admission: results from The Intensive Care Over Nations audit. Crit Care. 2018 Aug 3;22(1):188. doi: 10.1186/s13054-018-2112-z. PMID 30075798
- [Result] Yunos NM, Kim IB, Bellomo R, Bailey M, Ho L, Story D, Gutteridge GA, Hart GK. The biochemical effects of restricting chloride-rich fluids in intensive care. Crit Care Med. 2011 Nov;39(11):2419-24. doi: 10.1097/CCM.0b013e31822571e5. PMID 21705897
- [Result] Suetrong B, Pisitsak C, Boyd JH, Russell JA, Walley KR. Hyperchloremia and moderate increase in serum chloride are associated with acute kidney injury in severe sepsis and septic shock patients. Crit Care. 2016 Oct 6;20(1):315. doi: 10.1186/s13054-016-1499-7. PMID 27716310
- [Result] Raghunathan K, Shaw A, Nathanson B, Sturmer T, Brookhart A, Stefan MS, Setoguchi S, Beadles C, Lindenauer PK. Association between the choice of IV crystalloid and in-hospital mortality among critically ill adults with sepsis*. Crit Care Med. 2014 Jul;42(7):1585-91. doi: 10.1097/CCM.0000000000000305. PMID 24674927
- [Result] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Result] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925